CLINICAL TRIAL: NCT03670290
Title: Clinical Outcomes of Analgesia Methods in Patients With Hip Fracture
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mustafa Azizoğlu, Assistant Proffessor, Mersin University
Other Study IDs: MEUANEST001
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Hip Fractures
Keywords: hip fracture; fascia iliaca compartment catheter; epidural catheter; delirium; postoperative complications
MeSH Terms: conditions — Hip Fractures; Delirium; Postoperative Complications | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group I will receive 30 ml of Bupivacaine 0.25% solution through the fascia iliaca compartment catheter. Catheter will be inserted with US.
  Interventions: Procedure: Fascia iliaca compartment catheter
- Group 2: Group II will receive, morphine 0.1 mg/ml via patient controlled analgesia pump. every pump will be set 1 mg dose morphine per use and 15 min lockout time.
  Interventions: Procedure: patient controlled analgesia
- Group 3: Group III will receive 10 ml of Bupivacaine 0.25% solution through the epidural catheter.
  Interventions: Procedure: epidural catheter

INTERVENTIONS:
Procedure: Fascia iliaca compartment catheter — Patient will evaluate and if VAS score >3, catheter will be inserted and 30 ml bupivacaine 0.25% will be applied after admission. Dose will be repeated VAS>3 or patient enounce pain.
  Groups: Group 1
Procedure: epidural catheter — Patient will evaluate and if VAS score >3, catheter will be inserted and 10 ml bupivacaine 0.25% will be applied after admission. Dose will be repeated VAS>3 or patient enounce pain.
  Groups: Group 3
Procedure: patient controlled analgesia — Patient will evaluate and if VAS score >3, patient controlled analgesia pump will be set 1mg morphine/15 min lockout.
  Groups: Group 2

SUMMARY:
The goal of this study is to determine of clinical outcomes of analgesia methods. The primary outcomes are opioid consumption, static and dynamic visual analog scale (VAS) scores. Secondary outcomes are occurrence of side effects.

DETAILED DESCRIPTION:
Hip fracture is one of the most serious consequences of falls in the elderly, with a mortality of 10% at one month and 30% at one year. Factors of associated with increased morbidity and mortality have been researched to prevent complications.

Pain has been associated with delirium and depression in hip fracture patients. Besides, narcotic drugs are also associated with some side effects such as delirium, postoperative nausea and vomiting (PONV ), cardiovascular and respiratory depression. These clinical problems are especially important in the elderly population.

Fascia iliaca compartment block (FICB) is one of the methods applied for postoperative analgesia, which is applied under the inguinal ligament and distributes between the femoral nerve and lateral femoral cutaneous nerve block by volumetric effect. Recently, studies have been published on hip fracture patients using pop up technique in emergency services. Although many studies have shown that FICB is effective in perioperative analgesia, the effects of this method on complications and mortality rate have not yet been investigated.

The primary objective is to compare morphine consumption and VAS scores in patients with hip fracture who treated with epidural catheter, fascia iliaca compartment catheter or patient controlled analgesia.

The secondary objective is to determine complications. The investigators hypothesize that FICB catheter will provide good pain control same as epidural catheter, and will decrease complications such as delirium and pain with less mortality rate.

Patients with pain in the hip fracture, will be evaluated after admission to the hospital and analgesic treatment will be applied to patients with Visual Analog Pain Scale (VAS) score 3 and above.

Patients will be divided into three groups; Group I will include patients with treated FICB catheter, Group II will include patients with treated patient controlled analgesia, Group III will include patients with treated epidural catheter,

Catheters will be placed with US visualization in Group I. A hyperechoic needle will be used (18 G 80 mm) for inserting catheter in Group I and III.

Group I will receive 30 ml of Bupivacaine 0.25% solution through the fascia iliaca compartment catheter.

Group II will receive, morphine 0.1 mg/ml via patient controlled analgesia pump. every pump will be set 1 mg dose morphine per use and 15 min lockout time.

Group III will receive 10 ml of Bupivacaine 0.25% solution through the epidural catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients without communication problems (delirium, hearing loss, language problems etc.)
* Patients who do not use regular analgesic medication for any chronic disease
* Patients without any neurological deficit at the lower extremity
* Patients without renal or hepatic dysfunction
* Patients without bleeding diathesis
* Patients with isolated femur fractures

Exclusion Criteria:

* Patients with communication problems
* Patients who use regular analgesic medication for any chronic disease
* Patients with neurological deficits in the lower extremity
* Patients with renal or hepatic dysfunction
* Patients with bleeding diathesis
* Patients with multiple trauma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will be performed from 01/12/2018 to 01/06/2019. It is estimated to each group includes 40 patient.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | From the beginning of treatment to discharge (Totally 5 days)
  All perioperative morphine consumption will be recoreded every 6 hours.
Visual analogue score | From admission to second postoperative day. (Totally 5 days)
  Mean visual analogue scores will be compared for 3 groups. VAS score will measured from 0 to 10. Higher values represent worse outcome.

SECONDARY OUTCOMES:
incidence of postoperative complications in 30 day post-surgery. | From end of surgery to Day 30 after surgery (totally 30 days)
  Patients will be monitored and every serious complication related with surgery including respiratory failure, hypotension, delirium, thromboembolism, nausea and vomiting will be recorded. These events will be measured as percentage (%)

OTHER OUTCOMES:
Anticoagulant medication status in the S-FICB group | First day (15 min)
  The use of anticoagulant drugs will be questioned and recorded in the S-FICB group

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Azizoglu, Study Director — Mersin University, Anesthesia and Reanimation Department
Locations (1):
- Mustafa AZİZOĞLU, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Every entered data could share to other researchers
Supporting Information: Study Protocol
Time Frame: After 01/03/2019
Access Criteria: Sharing access will be depends on requests.